CLINICAL TRIAL: NCT03846856
Title: The IGF Axis Involvement in Immune Tumor Microenvironment in Ovarian Cancer and Its Clinical Significance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0080-18
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian cancer patients: Biopsy will be taken from ovarian cancer patients and sent to laboratory for analysis
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Biopsy taken during surgical procedure

SUMMARY:
The aim of this study is to evaluate the insulin-like growth factor (IGF) axis involvement in the immune tumor microenvironment in ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with epithelium ovarian cancer who have undergone surgery

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients diagnosed with epithelium ovarian cancer who have undergone or who plan to undergo surgery
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Involvement of IGF Axis in Ovarian Cancer | Two years
  Ovarian cancer specimens taken during surgical procedures will be evaluated and analyzed by flow cytometry assays to determine the involvement of the IGF axis in the immune tumor microenvironment in ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Bruchim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No